CLINICAL TRIAL: NCT06140004
Title: Investigating the Impact of Person-Centered Home-Based Palliative Care on Providers
Brief Title: Home-Based Palliative Care Impact on Providers
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Alexis Coulourides Kogan, PhD, Assistant Professor, University of Southern California
Other Study IDs: HS-17-00279; 1K99AG052647-01 (NIH); 5K99AG052647-02 (NIH); 4R00AG052647-03 (NIH); 5R00AG052647-04 (NIH)
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Palliative Care; Health Personnel
Keywords: Home-based palliative care; Healthcare providers; Qualitative methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HBPC Site 1: Northern/East California: This site implemented an evidence-based model of HBPC that consists of home visits by a trained, interdisciplinary palliative care team composed of a physician, nurse, social worker, and spiritual counselor. At this site, this core team was housed in an independent hospice agency and was also convened in-house by the ACO contract or MA plan. The insurance provider contracts with the core team, using a per member per month payment for patients enrolled in HBPC. The core team will provide pain and symptom management, psychosocial support, advanced care planning, disease management education, spiritual counseling, grief counseling, and other services in response to patient and caregiver needs. HBPC patients and their caregivers also will have access to a 24/7 helpline.
- HBPC Site 2: Northern/West California: This site implemented an evidence-based model of HBPC that consists of home visits by a trained, interdisciplinary palliative care team composed of a physician, nurse, social worker, and spiritual counselor. At this site, this core team was housed in an independent hospice agency and was also convened in-house by the ACO contract or MA plan. The insurance provider contracts with the core team, using a per member per month payment for patients enrolled in HBPC. The core team will provide pain and symptom management, psychosocial support, advanced care planning, disease management education, spiritual counseling, grief counseling, and other services in response to patient and caregiver needs. HBPC patients and their caregivers also will have access to a 24/7 helpline.
- HBPC Site 3: Southern California: This site implemented an evidence-based model of HBPC that consists of home visits by a trained, interdisciplinary palliative care team composed of a physician, nurse, social worker, and spiritual counselor. At this site, this core team was housed in an independent hospice and home health agency and was also convened in-house by the ACO contract or MA plan. The insurance provider contracts with the core team, using a per member per month payment for patients enrolled in HBPC. The core team will provide pain and symptom management, psychosocial support, advanced care planning, disease management education, spiritual counseling, grief counseling, and other services in response to patient and caregiver needs. HBPC patients and their caregivers also will have access to a 24/7 helpline.

SUMMARY:
This research challenges our current approach to fee-for-service palliative care and is significant because it will advance the fields of palliative and person-centered care, clinical practice, public policy, and health care financing. However, the most important effect will be on seriously ill patients and their families through increased access to palliative care outside of hospitals, enhanced palliative continuity across health settings, and improved affordability via reformed payment structures. Nation-wide replication of reimbursable HBCP models is anticipated.

DETAILED DESCRIPTION:
This study will undertake an effort to address the two-pronged gap in providing palliative care in the U.S. (episodic care and misaligned financing structures). This will be done by implementing an evidence-based Home-Based Palliative Care (HBPC) model-originally developed in managed care-into primary fee-for-service as a covered health benefit; the very first translation of this model by a private health insurer in the U.S. The purpose of the present study is to investigate the provider and organizational-level impact of implementing reimbursable HBPC in primary care with the goal of characterizing a set of implementation strategies and eliciting key mechanisms on how to widely replicate person-centered, reimbursable HBPC in primary care settings across the country. To this end, seven research questions will be answered that address the study purpose pertaining to feasibility, barriers, facilitators, person-centeredness, and job satisfaction. This study is guided by the Diffusion of Innovations theory. The investigators will conduct primary collection and analysis of qualitative focus group data at each study site. Key outcomes for the qualitative component include feasibility, barriers, and facilitators of translating HBPC, as well as characteristics associated with rate of HBPC diffusion and implementation strategies. This project challenges our current approach to fee-for-service palliative care and seeks to shift current research. Nation-wide replication of reimbursable HBCP models is anticipated.

ELIGIBILITY:
Inclusion Criteria:

• Current member of the Home-Based Palliative Care (HBPC) team or organization's leadership team

Exclusion Criteria:

* No interaction with palliative care patients or palliative care arm of organization
* Unable to speak and read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participant were members of the HBPC service at each organization. The investigators sought participants with a wide variety of disciplines, roles, and experiences. This included targeting frontline providers consistent with the core clinical team outlined in the HBPC model (i.e., physician, nurse [RNs], social worker [LCSWs, MSWs], and chaplain), in addition to other site team members such as advance practice providers (NPs, PAs), patient coordinators/liaisons, admissions assistants, and leadership.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Confidence in Team | 12-months
  Self-reported rating of confidence in HBPC team to implement the intervention as stated, on a scale of 1-10 (1=not confident at all; 10=extremely confident)

SECONDARY OUTCOMES:
Confidence in Self | 12-months
  Self-reported rating of confidence in self to implement the intervention as stated, on a scale of 1-10 (1=not confident at all; 10=extremely confident)

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Coulourides Kogan, PhD, Principal Investigator — University of Southern California
Locations (3):
- United States (3):
  - By the Bay Health, Larkspur, California
  - Snowline Hospice, Sacramento, California
  - HavenHealth, Signal Hill, California

IPD SHARING:
Plan to Share IPD: No
De-identified IPD in the form of focus groups transcripts and demographic survey data will be shared upon request. Legitimate requests by researchers can be made in writing directly to the study PI.